CLINICAL TRIAL: NCT03093194
Title: Vaginal Antimicrobacterial Preparation Before Cesarean Secation for Endometritis Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, HILA BEN-ASHER MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RAMBAMMV
Record Dates: First submitted 2017-03-12; First posted 2017-03-28 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: A Known Allergy to Antiseptic Soap; Women Who Had Any Infection in the Perioperative Period; A Known Allergy to Chlorohexidine Alcohol or Shellfis

STUDY DESIGN:
Intervention Model Description: Patients will be randomaly assigned into two groups. The experiment group will not undergo vaginal preparation. The control will undergo perioperative vaginal preparation with antiseptic soap and chlorohexidine-alcohol.
  All patients participating in this trail will sign a written informed consent. All patients will receive preventative antibiotics peri-operatively according to the our hospital protocol.
  Exclusion criteria are a known allergy to antiseptic soap, chlorohexidine-alcohol or shellfish, or patients who had any infection in the perioperative period.
  Inclusion criteria: an elective or emergent CS in a woman who did not report having a fever or skin infection signs in the 5 days prior to surgery.
  Once a patient is admitted to the delivery room, approximately 7 days to several hours before CS each patient will be assigned randomly to a group using a computerized randomization software.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The study is not double blind, therefore is subjected to the care provider bias. Outcomes assessment might also be over or under evaluated by the physician following the patients outside the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women going CS without vaginal preparation before surgery (Active Comparator): Women going CS without vaginal preparation before surgery. No vaginal preparation before CS with Septal soap and septol.
  Interventions: Other: No vaginal preparation before CS with Septal soap and septol.
- Women going CS with vaginal preparation before surgery (Placebo Comparator): Women going CS with vaginal preparation before surgery. vaginal preparation before CS with Septal soap and septol.
  Interventions: Other: vaginal preparation before CS with Septal soap and septol.

INTERVENTIONS:
Other: vaginal preparation before CS with Septal soap and septol. — vaginal preparation before CS with Septal soap and septol.
  Arms: Women going CS with vaginal preparation before surgery
Other: No vaginal preparation before CS with Septal soap and septol. — No vaginal preparation before CS with Septal soap and septol.
  Arms: Women going CS without vaginal preparation before surgery

SUMMARY:
The investigators designed a randomized controlled trial to evaluate whether perioperative Vaginal preparation is superior to no Vaginal preparation in decreasing post CS endometritis. Since CS is performed in about 30% of all births and infection complicates 6-11% of all CS reducing the rate of this post CS complication can have a major impact not only on the hospital occupancy and costs but also on the new mother experience and ability to face the challenge that awaits for her with her newborn.

In this study patients will be randomly assigned into two groups. The experiment group will not undergo any vaginal preparation. The control will undergo perioperative vaginal preparation with antiseptic soap followed by chlorohexidine-alcohol Both groups will be checked for cervical dilation with sterile gloves before surgery.

Primary outcome - signs of endometritis (e.g. erythema around surgical scar, discharge or pain). Patients will be followed daily until discharge. A blood count will be drewn before discharge to rule out signs of infection. Patients will be contacted 6 weeks after surgery by telephone to inquire about any signs of infection, Emergency Room visits or ambulatory visits to the doctor due to endometritis. The participants will be asked if they had positive skin culture or other wound complications such as cellulitis, seroma or scar separation.

The investigators estimated that 1040 patients will have to enroll into the study, 520 in each group in order to have 80% power to detect 50% difference in the endometritis rates between the two groups with a two tailed α level of 0.05.

The data analysis was conducted according to the per-protocol principle.

DETAILED DESCRIPTION:
BACKGROUND In the last decades, caesarean sections rate have escalated steadily worldwide. In 2013, more than 32.7% births in the United States were by cesarean section 1. These high rates of cesarean deliveries are of substantial concern due to the potential associated complications such as endometritis (6-11%) 2, wound complications (1-2%) 2, hemorrhage, injury to pelvic organs (0.2-0.5%)2, and thromboembolic disorders (100-240 per100,000) 3 .

One of the common complications following CS is endometritis. Post cs endometritis prolongs the patient hospitalization therefore not only elevating the hospital's costs but also intervening with the mother's ability to take care and bond with the new baby. It also poses a risk on future fertility by increasing the risk of long term complications including Asherman's syndrome and in rare cases may necessitate a hysterectomy. Therefore, decreasing post cs endometritis is a substantial goal for the OBGYN practitioner.

In the current literature a debate surrounds the contribution of perioperative vaginal preparation to the prevention of post CS endometritis. In a meta-analysis of seven randomized trials vaginal preparation before CS using povidone-iodine in addition to abdominal preparation showed a significantly reduced frequency of postoperative endometritis 4. However, this benefit was restricted to women with ruptured membranes and the benefit for all women undergoing CS is still undetermined. Currently there is no recommendation for routine perioperative vaginal preparation before CS.The benefit of perioperative vaginal preparation is the motivation for this study. The design of this study is a randomized controlled trial meant to evaluate whether perioperative Vaginal preparation is superior to no Vaginal preparation in decreasing post CS endometritis Furthermore, in past settings povidone-iodine had been tested. Povidone-iodine compromised the thyroid function of the physicians and was replaced by chlorohexdine solution. Since that transition no trails have revised the prevention of endometritis after vaginal preparation with chlorhexidine.

Since CS is performed in about 30% of all births and infection complicates 6-11% of all CS reducing the rate of this post CS complication can have a major impact not only on the hospital occupancy and costs but also on the new mother experience and ability to face the challenge that awaits for her with her newborn.

METHODS Women will be randomly assign the patients into two groups. The experiment group will not undergo any vaginal preparation. The control will undergo perioperative vaginal preparation with antiseptic soap followed by chlorohexidine-alcohol. Both groups will be checked for cervical dilation with sterile gloves before surgery.

All patients participating in this trail will sign a written informed consent. All patients will receive preventative antibiotics peri-operatively according to the our hospital protocol.

Exclusion criteria are a known allergy to antiseptic soap, chlorohexidine-alcohol or shellfish, or patient who had any infection in the perioperative period.

Inclusion criteria: an elective or emergent CS in a patient who did not report having a fever or skin infection signs in the 5 days prior to surgery.

Once a patient is admitted to the delivery room, approximately 7 days to several hours before the decision to perform a CS will be made and all inclusion criteria met, each patient will be assigned randomly to a group using a computerized randomization software.

Primary outcome - signs of endometritis (e.g. erythema around surgical scar, discharge or pain). Patients will be followed daily until discharge. A blood count will be drewn before discharge to rule out signs of infection. Patients will be contacted 6 weeks after surgery by telephone to inquire about any signs of infection, Emergency Room visits or ambulatory visits to the doctor due to endometritis. The participants will be asked if they had positive skin culture or other wound complications such as cellulitis, seroma or scar separation.

STATISTICAL ANALYSIS The sample size was calculated for this trail assuming a rate of endometritis of 6% on the basis of the rates known in literature 2 . A 4% lower rate of endometritis is expected in the vaginal preparation group compared with the no vaginal preparation group. A total of 1040 patients will have to enroll in our study, 520 in each group in order to have 80% power to detect 50% difference in the endometritis rates between the two groups with a two tailed α level of 0.05.

The data analysis was conducted according to the per-protocol principle. Data will be stratified according to other factors such as maternal age, BMI, medical background and specifically diabetes or autoimmune conditions, gestational age, and ethnicity. Relative risk of primary outcome will be calculated with 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

an elective or emergent CS in a woman who did not report having a fever or skin infection signs in the 5 days prior to surgery.

Exclusion Criteria:

1. a known allergy to antiseptic soap, chlorohexidine-alcohol or shellfish
2. women who had any infection in the perioperative period.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2017-04-10 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
rates of endometritis | 2.5 years
  rates of endometritis

SECONDARY OUTCOMES:
rates of Urinary Tract Infections | 2.5 years
  rates of Urinary Tract Infections

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895